CLINICAL TRIAL: NCT01041664
Title: Bad Genes or Genes Behaving Badly
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Krista Casazza, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F091006003
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Body Composition; Energy Balance; Metabolism
Keywords: nutrigenomics; admixture; Hispanic American; body composition; Association of diet and body composition; Association between genes and body composition; Association between gen by diet interaction and body composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples will be labeled with the study protocol number, a unique identifier, and the date of collection.
  Specimens will be obtained by the nursing staff at the PCIR. The PCIR processing lab will process the samples, which will then be stored in a locked freezer at -80oC in the restricted access CNRU Metabolism Core lab (WEBB 337).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A key factor in the determination of body composition over the lifecourse is fat accumulation during childhood. Periods of life associated with the greatest changes in organ development and growth, i.e. early childhood, have the most significant effect on body composition, energy balance, and metabolism. Early childhood (age 3 to 7 years) represents a critical transition for the basis of adaptability in body composition, due to the rapid growth and development that occurs. Plausibly the phenotype underlying obesity and related health risk may be determined by body composition during this critical period.

Our previous research in children has consistently indicated that HA children accumulate greater amounts of fat, particularly in the intra-abdominal compartment, even at similar a BMI, and lower bone mineral content relative to EA children. The reason for these differences in body composition over the lifecourse is not clear.

Racial/ethnic differences in risk factors for health, including 'thriftiness' in body fat accumulation are often evident before the age of 7, suggesting that the racial/ethnic differences in energy utilization and subsequent fat storage may be accounted for by genetic make-up, the environment (e.g. diet), or an interaction of the two. The physiologic or behavioral process(es) that cause(s) certain children to take a trajectory towards obesity while others accrue less fat is not known. However, the economic decision of fuel utilization is a physiologic trait enabling the body to choose between shuttling 'energy' towards accrual of a particular tissue (e.g. bone vs. fat) and this trait likely has a genetic component. This genetic component may be embedded in fat storage capacity evolved from gene by environment interactions that promote thrift, particularly conserved in some populations. Although genetic background plays a role, it not known whether there is a relationship between genetic background, known candidate genes or candidate pathways and environmental contributors (e.g. diet) that impact body composition trajectory. Of central importance to our understanding of early fat mass accumulation in health disparities are the mechanisms that lead to chronic disease progression.

It is likely that variations within candidate genes may have a differential impact on individuals based on their genetic background. It is also probable that body composition is influenced by many genes, often within the same metabolic pathways, with small individual effects. These genes may not be significantly associated individually, but when examined as a unit (in a candidate pathway or gene-gene interaction framework) the association becomes significant. Further, children's early environmental exposures (e.g. diet) may interact with both genetic background and variations in candidate genes along resulting in alterations in body composition that predispose HA to excess fat accumulation throughout the lifecourse. To that end, the following specific aims will be evaluated:

Aim 1. To examine the associations between genetic admixture and body composition in children aged 3-7 years after controlling for dietary intake.

1. Hypothesis 1.1: There is a direct association between Amerindian admixture and fat mass and in inverse association between Amerindian admixture and bone mass.
2. Hypothesis 1.2: There is a direct association between energy intake and fat accumulation and the relationship will be particularly evident in individuals with a greater proportion of Amerindian admixture.

Aim 2. To examine the associations between genetic admixture and bone marrow fat in children aged 3-7 years after controlling for dietary intake.

1. Hypothesis 2.1: There is a direct association between Amerindian admixture and bone marrow fat.
2. Hypothesis 2.2: There is a direct association between energy intake and fat accumulation in bone marrow and the relationship will be particularly evident in individuals with a greater proportion of Amerindian admixture.

Aim 3. To examine the relationship between variation in candidate genes and pathways and Amerindian admixture controlling for dietary intake.

a. Hypothesis 3.1: Amerindian admixture will be associated with variations in candidate genes and pathways known to be associated with fat accumulation.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Hispanic American
* Healthy, not under the care of a doctor
* Not taking medications known to affect body composition or metabolism

Exclusion Criteria:

* Not meeting above criteria

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be healthy children self-identifed as Hispanic American aged 3 to seven years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of diet by gene interactions on body composition measures in Hispanic American children | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States